CLINICAL TRIAL: NCT02170155
Title: MRI-changes in Morphometry and Cerebro Spinale Fluid (CSF) Flow in Spinal Cord Disorders
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Foundation Wings For Life (Other); Balgrist Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-2012-0343/PB_2016-00623
Record Dates: First submitted 2014-06-05; First posted 2014-06-23 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Spinal Injury
MeSH Terms: conditions — Spinal Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Patients with CSM
- Patients with spinal injury (SCI)
- Healthy controls

SUMMARY:
Understanding the onset and progression of spinal cord disorders is an important aim in clinical neurology. An early diagnosis with consequent therapy might prevent the progression of disability. Therefore, we aim to determine structural and dynamic changes in the microstructure of the spinal cord and CSF, and to explore the relationships between the MRI parameters, clinical disability, and electrophysiology.

In some patients that undergo decompressive surgery CSF pressure will be measured invasive perioperative for 24h to find out if functional limitations and structural changes correlate with the spinal pressure and the spinal perfusion when the spinal cord is damaged.

ELIGIBILITY:
Inclusion Criteria:

* Cervical injury
* Informed consent
* Age 18-80
* CSM

Exclusion Criteria:

* No other neurologic disorder and psychiatric disorder
* Seizure
* MRI incompatibility
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with spinal cord disorder and CSM
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2012-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Morphometric changes and changes in cerebro spinal fluid (CSF) flow and spinal cord movement in patients and control subjects will be correlated to functional deficits and neurophysiological data (regression model analysis). | Each patient will undergo a MRI scan, clinical and electrophysiological examinations at baseline, after 6 months and after 1, 2, 3, 4, and 5 years. Controls will undergo 1 MRI scan and some scan of retest analysis
Assessment of CSF pressure dynamics in the perioperative setting | Perioperative for 24hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Pfender N, Jutzeler CR, Hubli M, Scheuren PS, Pfyffer D, Zipser CM, Rosner J, Friedl S, Sutter R, Spirig JM, Betz M, Schubert M, Seif M, Freund P, Farshad M, Curt A, Hupp M. Potential thresholds of critically increased cardiac-related spinal cord motion in degenerative cervical myelopathy. Front Neurol. 2024 Jun 24;15:1411182. doi: 10.3389/fneur.2024.1411182. eCollection 2024. PMID 38978814
- [Derived] Kheram N, Boraschi A, Pfender N, Spiegelberg A, Kurtcuoglu V, Curt A, Schubert M, Zipser CM. Queckenstedt's test repurposed for the quantitative assessment of the cerebrospinal fluid pulsatility curve. Acta Neurochir (Wien). 2023 Jun;165(6):1533-1543. doi: 10.1007/s00701-023-05583-w. Epub 2023 Apr 20. PMID 37079108
- [Derived] Zipser CM, Pfender N, Spirig JM, Betz M, Aguirre J, Hupp M, Farshad M, Curt A, Schubert M. Study protocol for an observational study of cerebrospinal fluid pressure in patients with degenerative cervical myelopathy undergoing surgical deCOMPression of the spinal CORD: the COMP-CORD study. BMJ Open. 2020 Sep 21;10(9):e037332. doi: 10.1136/bmjopen-2020-037332. PMID 32958488